CLINICAL TRIAL: NCT06521060
Title: The Role of Pre-Surgical Tru - Cut Biopsy in the Management of Atypical Myometrial Lesions
Acronym: MYSTR
Status: Not yet recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Sponsor
Other Study IDs: NW24J-03-00025
Record Dates: First submitted 2023-12-03; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2023-11

CONDITIONS: Leiomyosarcoma
Keywords: tru cut biopsy; leiomyoma
MeSH Terms: conditions — Leiomyosarcoma; Leiomyoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Following samples will be stored in biobanks at each respective institution: tumor sample DNA (isolated from one snap-frozen TCB sample); representative formalin-fixed paraffin-embedded (FFPE) tumor tissue block and representative FFPE non-tumor myometrial tissue block (both harvested during curative surgery). All samples will be collected with the intention to be used for future translational and exploratory research, including studies that aim to evaluate the association between biomarkers and clinical-surgical-pathological characteristics. All samples will be stored in the biobank at the respective institution.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tru cut biopsy: A single arm, prospective, multicentric cohort study. A total of 250 patients is planned to be enrolled, accounting for an estimated 15% dropout rate.
  Interventions: Procedure: tru cut biopsy

INTERVENTIONS:
Procedure: tru cut biopsy — Proving that preoperative TCB could provide accurate information about the histological nature of the tumor would have great impact for setting an adequate, tailored, oncologically safe treatment approach.

SUMMARY:
The Tru-cut biopsy (TCB) for targeting pelvic tumors is well established in gynecologic oncology. However, its reliability for differentiating of uterine sarcoma in "myoma-like" uterine lesions has been confirmed by only a few studies, which were either retrospective or provided only pilot result on the limited number of prospectively enrolled patients (N=34). Proving that preoperative TCB can provide accurate information about the histological nature of the tumor would have great impact for setting an adequate tailored oncologically safe approach, especially in patients with sonographically atypical lesions. Additionally, the biopsy should be safe, with transcervical, transuterine cavity ("in organ" biopsy) approaches preferred to avoid the risk of needle canal contamination if sarcoma is diagnosed. The purpose of this study is to evaluate the accuracy of the Tru-cut biopsy (TCB) of sonographically atypical myometrial lesions as a complementary diagnostic method in the preoperative management of patients scheduled for uterus preserving procedure or hysterectomy. Additionally, we aim to assess the impact of this procedure on patients´ quality of life and clinical management. MYSTR is a single arm, prospective, multicentric cohort study.

DETAILED DESCRIPTION:
A total of 250 patients is planned to be enrolled, accounting for an estimated 15% dropout rate. Study data will be collected and managed using REDCap (Research Electronic Data Capture) open-source platform, which allows for the secure collection of research data via a web-based interface. REDCap was developed by Vanderbilt University in Nashville, Tennessee, is used by Charles University in Prague under a standing agreement to allow the usage of REDCap for academic and research purposes. The REDCap platform environment is compliant with 21 CFR Part 11, FISMA, HIPAA, and GDPR.

Patients will be identified at each of the participating site. If a patient meets all inclusion criteria, she will be informed about the study and asked to sign an informed consent (ICF). All patients referred for TCB will have their blood count and baseline coagulation parameters checked prior to performing the biopsy to eliminate bleeding complications. All patients will undergo a standard-of-care ultrasound examination with a focus on the description of the fibroid with atypical features according to the MUSA statement and/or Basel sarcoma scale score (BSS). A patient will be included in the study if she will meet one or more of the following MUSA criterion: irregular tumor borders, cystic areas in the lesion (as a sign of central necrosis), nonuniform echogenicity, moderate-to-abundant intralesional vascularity and an absence of calcifications, and/or BSS total score ≥ 1.

The patient will be further referred to MRI imaging (optional) and will undergo TCB within 4 weeks after US exam. In selected centers which will decide to participate in this optional part of the trial, all patients with ≥ 1 MUSA criterion and/or BSS total score ≥ 1 based on the US examination will be referred for MRI imaging. Images will be acquired with 3T MRI. The sequences parameters (Sagittal T2, Coronal T2, Axial T2, Axial DWI, Axial T1 3D DIXON, Axial Perfusion T1 3D, Axial T1 3D DIXON post contrast) will be evaluated in accordance with European Society of Urogenital Radiology (ESUR) guidelines. Two experienced readers in gynecologic oncology imaging will review all MRI images and calculate the MRI score.

The tru-cut biopsy is performed as an out-patient procedure without the need of any anesthesia in lithotomic position. Using an automatic biopsy gun and 18-gauge disposable core tissue biopsy needle four tissue cylinder samples are taken from the tumor. If the localization of the lesion and anatomical conditions allow, the transcervical approach without breaking the continuity of the perimetrium is preferred. If the lesion is localized in the uterine doom, or targetable by the uterine cavity, the transcervical canal approach is feasible and should be considered. If both above-described methods are not feasible, a transvaginal approach is also possible. In all cases transvaginal US is used for correct navigation. Patients will be observed for 30 minutes following the biopsy and then discharged. Other follow up of the patients will be done 24 hours and two weeks after the procedure via phone with the assessment of the patient´s pain, overall experience, and eventual complications.

Intraoperative and early post-procedural complications will be evaluated, and adverse events will be assessed on the 14th post-TCB day according to the Clavien-Dindo Surgical complications classification. Pain will be assessed during the TCB, 30 minutes after the procedure, and after 24 hours using the Numeric rating scale (NRS). Overall experience will be assessed using questionnaire: FACIT-TS-G (Version 4) 30 minutes after the procedure.

Specimen evaluation will be conducted at each participating site by dedicated, experienced pathologist according to standard diagnostic procedures. The biological nature of spindle cell leiomyocellular tumors will be determined according to Table 2 (modified from the WHO classification of female genital tumors 2020).

If necessary, immunohistochemical or molecular examination will be used. For smooth muscle lesions the gene mutation status of PTEN, pRb, TP53, MTAP, ATRX, and DAXX will be analyzed. In lesions of other histological types, RNA next-generation sequencing will be performed, optionally accompanied by immunohistochemical examination. These examinations are routinely performed as a part of standardized diagnostic procedures and will not be covered by the project's expenses. Histology findings from other than the main sight that will fail to meet the characteristics of conventional leiomyoma (either from TCB or definitive histology result) will undergo a second evaluation at the main site by a senior gyneco-pathologist. Following samples will be stored in biobanks at each respective institution: tumor sample DNA (isolated from one snap-frozen TCB sample); representative formalin-fixed paraffin-embedded (FFPE) tumor tissue block and representative FFPE non-tumor myometrial tissue block (both harvested during curative surgery). All samples will be collected with the intention to be used for future translational and exploratory research, including studies that aim to evaluate the association between biomarkers and clinical-surgical-pathological characteristics. All samples will be stored in the biobank at the respective institution. Participation in the translatory part is not obligatory for the trial participation but is highly recommended. A separate consent form will be provided to the patient to obtain permission for all biological material storage and future translational studies. Based on the histology result obtained from the TCB, patients will be categorized into three groups. Subsequent clinical management will be determined according to the appropriate group:

Subgroup 1: Patients with a typical benign histological result of TCB will undergo elective surgery within 8 weeks from receiving the results, with a preference of a minimally invasive approach, i.e., most often laparoscopic myomectomy or laparoscopic hysterectomy.

Subgroup 2: Patients with an atypical histological result of TCB (i.e., other than conventional leiomyoma but with no signs of malignancy) will undergo elective surgery within 6 weeks from receiving the results, with a preference of laparoscopy but excluding unprotected power morcellation of pathological tissue.

Uncontained morcellation will be used strictly for tumors with benign TCB histology and nonsuspicious perioperative appearance of resected uterine tumor. Contained morcellation technique will be strictly preferred for all other tumors, i.e., with non-standard TCB histology and/or atypical or suspicious perioperative appearance, or standard TCB histology and atypical or suspicious perioperative appearance.

Subgroup 3: Patients with a histological result from the TCB that are clearly malignant or suspicious for malignancy undergo open surgery, specifically abdominal hysterectomy. In cases of women with incomplete reproductive plans, open resection of the tumor may be performed after detailed consultation with the oncogynecological team and the patient, a secondary hysterectomy may be added based on the result of definitive histology. The procedure should be done as soon as possible, with a maximum interval between the result of TCB histology and elective surgery no more than 3 weeks.

In cases of tumors without penetration through the uterine serosa (according to US and perioperatively) and without requiring morcellation for the specimen evacuation, total laparoscopic hysterectomy can be performed.

Subgroup 4: In case of invalid TCB histology result, the patient will undergo contained morcellation during laparoscopic procedure or open surgery within 4 weeks after the TCB.

The definitive histology results from the surgery will be evaluated using the same histopathological criteria as in TCB histology. Definitive histology will be compared with the histological results from the pre-surgical TCB.

For the primary endpoint analysis, the accuracy of the histological results from TCB will be established using the definitive postoperative histological results as a reference standard.

The sample size of 217 patients with sonographically atypical myometrial lesions was calculated to establish the accuracy of the diagnostic method, with the degree of estimate precision of 0.07, 95% confidence and 80% power; assuming ratio between patients with/ without atypical lesion as per final pathology of 23:77, as based on the retrospective database data. Considering a possible dropout or unavailability of data in 15% of the patients, the final sample size reaches 250 patients. Analysis was computed using PASS 13 Power Analysis and Sample Size Software (2014). NCSS, LLC. Kaysville, Utah, USA, ncss.com/software/pass.

If this trial proves the accuracy of TCB of myometrial lesion, it could provide a new diagnostic tool and significantly impact the clinical practice.

A positive study outcome could establish level A evidence for a change of international standards and implement prehabilitation into a routine clinical practice. On a national level, the study aims to standardize and improve the care for gynecological patients with sonographic atypical myometrial lesions. A primary endpoint final analysis is intended for publication in a top medical journal. The study could also provide prospective genomic characterization analyses of myometrial tumors as well as the exploratory analysis of the reliability of individual imaging methods in the preliminary selection of patients with atypical myometrial findings.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age ≥ 18 years
* Women indicated for uterus-preserving surgery (tumour resection) or hysterectomy for myometrial lesion ('myoma-like' uterine tumour(s))
* USG finding of atypical myometrial lesion/s a

Exclusion Criteria:

patient 's refusal

* age < 18 years
* ongoing pregnancy
* inability to perform TCB /contraindications for TCB (trombocytopenia, coagulopathy, PID, colpitis) or definitive surgery (myomectomy or hysterectomy)
* USG finding of more than 2 atypical lesion/s with a diameter ≤ 20 mm and ≥ 100 mm
* inability to perform any of the 3 core needle biopsy approaches (transvervical, trans uterine cavity, transvaginal) because of anatomical, localization issues. The percutaneous transabdominal biopsy is not allowed
* Polymyomatous uterus that may not be examined adequately with routine transvaginal ultrasound
* myoma (which would be subject to TCB) type 7 according to FIGO classification 16
* history of conservative hormonal therapy less than 3 months prior to study enrolment
* history of conservative therapy via uterine artery embolisation or laparoscopic uterine artery occlusion
* history of pregnancy less than one year prior to study enrollment

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Age ≥ 18 years
  * Women indicated for uterus-preserving surgery (tumour resection) or hysterectomy for myometrial lesion ('myoma-like' uterine tumour(s))
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Rate of accuracy | 3 years
  Accuracy is defined as the concordance of the results of preoperative histology from TCB with the result of definitive histology from the operative specimen

SECONDARY OUTCOMES:
Rate of adequately performed TCBs | 3 years
  defined as the number of TCBs with adequate encroachment of the lesion with bioptic needle (by the US) and sufficient tissue sample for the histopathological analysis to the total number of TCBs.
Number of complications | 3 years
  number of complications after TCB divided by the number of patients. Intraoperative and early post-procedural complications will be assessed using a questionnaire. Adverse events will be assessed 14th post-TCB day according to the Clavien-Dindo Surgical complications classification
Pain associated with TCB | 24 hours
  Assessment of patient´s pain during, 30 minutes after, and 24 hours after the procedure using the Numeric rating scale (NRS)
Comparison of the preoperative MRI examination to US imaging | 3 years
  Testing the superiority of either approach, sensitivity and specificity of the MRI imaging when compared to US examination will be analyzed
Patient satisfaction with the diagnostic MRI and TCB | 3 years
  1 questionnaire: Patient experience of the diagnostic modalities will be assessed using developed and validated Patient Satisfaction Questionnaire
Impact of TCB on clinical management | 3 years
  the change of clinical management of patients with uterine "myoma-like" tumors caused by the TCB histology results (frequency of open surgeries and rate of necessary use of contained morcellation during laparoscopic myomectomy or hysterectomy)
Frequency of non-standard histological findings | 3 years
  the frequency of atypical histological findings (other than conventional leiomyoma) from the results of definitive histology in the group of women with sonographically atypical initial findings
Validation of the US markers of atypical myometrial lesions | 3 years
  External validation of the MUSA statement and/or Basel sarcoma scale score (BSS), correlation of respective imaging score and final pathology result

CONTACTS AND LOCATIONS:
Overall Officials: Kristyna Hlinecka, Principal Investigator — Charles University, Czech Republic
Locations (1):
- General hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abdel Wahab C, Jannot AS, Bonaffini PA, Bourillon C, Cornou C, Lefrere-Belda MA, Bats AS, Thomassin-Naggara I, Bellucci A, Reinhold C, Fournier LS. Diagnostic Algorithm to Differentiate Benign Atypical Leiomyomas from Malignant Uterine Sarcomas with Diffusion-weighted MRI. Radiology. 2020 Nov;297(2):361-371. doi: 10.1148/radiol.2020191658. Epub 2020 Sep 15. PMID 32930650
- [Background] Bonneau C, Thomassin-Naggara I, Dechoux S, Cortez A, Darai E, Rouzier R. Value of ultrasonography and magnetic resonance imaging for the characterization of uterine mesenchymal tumors. Acta Obstet Gynecol Scand. 2014 Mar;93(3):261-8. doi: 10.1111/aogs.12325. PMID 24372487
- [Background] Kubik-Huch RA, Weston M, Nougaret S, Leonhardt H, Thomassin-Naggara I, Horta M, Cunha TM, Maciel C, Rockall A, Forstner R. European Society of Urogenital Radiology (ESUR) Guidelines: MR Imaging of Leiomyomas. Eur Radiol. 2018 Aug;28(8):3125-3137. doi: 10.1007/s00330-017-5157-5. Epub 2018 Feb 28. PMID 29492599
- [Background] Kawamura N, Ichimura T, Ito F, Shibata S, Takahashi K, Tsujimura A, Ishiko O, Haba T, Wakasa K, Ogita S. Transcervical needle biopsy for the differential diagnosis between uterine sarcoma and leiomyoma. Cancer. 2002 Mar 15;94(6):1713-20. doi: 10.1002/cncr.10382. PMID 11920533
- [Background] Tamura R, Kashima K, Asatani M, Nishino K, Nishikawa N, Sekine M, Serikawa T, Enomoto T. Preoperative ultrasound-guided needle biopsy of 63 uterine tumors having high signal intensity upon T2-weighted magnetic resonance imaging. Int J Gynecol Cancer. 2014 Jul;24(6):1042-7. doi: 10.1097/IGC.0000000000000189. PMID 24927248
- [Background] Verschuere H, Froyman W, Van den Bosch T, Van Hoefs M, Kaijser J, Van Schoubroeck D, Van Rompuy AS, Vergote I, Timmerman D. Safety and efficiency of performing transvaginal ultrasound-guided tru-cut biopsy for pelvic masses. Gynecol Oncol. 2021 Jun;161(3):845-851. doi: 10.1016/j.ygyno.2021.03.026. Epub 2021 Apr 12. PMID 33858675
- [Background] Mascilini F, Quagliozzi L, Moro F, Moruzzi MC, De Blasis I, Paris V, Scambia G, Fagotti A, Testa AC. Role of transvaginal ultrasound-guided biopsy in gynecology. Int J Gynecol Cancer. 2020 Jan;30(1):128-132. doi: 10.1136/ijgc-2019-000734. Epub 2019 Oct 23. PMID 31645428
- [Background] Wang L, Li S, Zhang Z, Jia J, Shan B. Prevalence and occult rates of uterine leiomyosarcoma. Medicine (Baltimore). 2020 Aug 14;99(33):e21766. doi: 10.1097/MD.0000000000021766. PMID 32872073
- [Background] Raffone A, Raimondo D, Neola D, Travaglino A, Giorgi M, Lazzeri L, De Laurentiis F, Carravetta C, Zupi E, Seracchioli R, Casadio P, Guida M. Diagnostic accuracy of MRI in the differential diagnosis between uterine leiomyomas and sarcomas: A systematic review and meta-analysis. Int J Gynaecol Obstet. 2024 Apr;165(1):22-33. doi: 10.1002/ijgo.15136. Epub 2023 Sep 21. PMID 37732472
- [Background] Knipprath-Meszaros AM, Tozzi A, Butenschon A, Reina H, Schoetzau A, Montavon C, Heinzelmann-Schwarz V, Manegold-Brauer G. High negative prediction for the Basel sarcoma score: Sonographic assessment of features suspicious of uterine sarcoma. Gynecol Oncol. 2023 Jul;174:182-189. doi: 10.1016/j.ygyno.2023.05.005. Epub 2023 May 19. PMID 37210928
- [Background] De Bruyn C, Ceusters J, Vanden Brande K, Timmerman S, Froyman W, Timmerman D, Van Rompuy AS, Coosemans A, Van den Bosch T. Ultrasound features using MUSA terms and definitions in uterine sarcoma and leiomyoma: cohort study. Ultrasound Obstet Gynecol. 2024 May;63(5):683-690. doi: 10.1002/uog.27535. Epub 2024 Apr 5. PMID 37970762
- [Background] Bell SW, Kempson RL, Hendrickson MR. Problematic uterine smooth muscle neoplasms. A clinicopathologic study of 213 cases. Am J Surg Pathol. 1994 Jun;18(6):535-58. PMID 8179071
- [Background] Bedient CE, Magrina JF, Noble BN, Kho RM. Comparison of robotic and laparoscopic myomectomy. Am J Obstet Gynecol. 2009 Dec;201(6):566.e1-5. doi: 10.1016/j.ajog.2009.05.049. Epub 2009 Aug 15. PMID 19683685
- [Background] Suzuki Y, Wada S, Nakajima A, Fukushi Y, Hayashi M, Matsuda T, Asano R, Sakurai Y, Noguchi H, Shinohara T, Sato C, Fujino T. Magnetic Resonance Imaging Grading System for Preoperative Diagnosis of Leiomyomas and Uterine Smooth Muscle Tumors. J Minim Invasive Gynecol. 2018 Mar-Apr;25(3):507-513. doi: 10.1016/j.jmig.2017.08.660. Epub 2017 Oct 24. PMID 29079462
- [Background] Cotrino I, Carosso A, Macchi C, Baima Poma C, Cosma S, Ribotta M, Viora E, Sciarrone A, Borella F, Zola P. Ultrasound and clinical characteristics of uterine smooth muscle tumors of uncertain malignant potential (STUMPs). Eur J Obstet Gynecol Reprod Biol. 2020 Aug;251:167-172. doi: 10.1016/j.ejogrb.2020.05.040. Epub 2020 May 25. PMID 32505056
- [Background] Ludovisi M, Moro F, Pasciuto T, Di Noi S, Giunchi S, Savelli L, Pascual MA, Sladkevicius P, Alcazar JL, Franchi D, Mancari R, Moruzzi MC, Jurkovic D, Chiappa V, Guerriero S, Exacoustos C, Epstein E, Fruhauf F, Fischerova D, Fruscio R, Ciccarone F, Zannoni GF, Scambia G, Valentin L, Testa AC. Imaging in gynecological disease (15): clinical and ultrasound characteristics of uterine sarcoma. Ultrasound Obstet Gynecol. 2019 Nov;54(5):676-687. doi: 10.1002/uog.20270. Epub 2019 Oct 7. PMID 30908820
- [Background] Van den Bosch T, Dueholm M, Leone FP, Valentin L, Rasmussen CK, Votino A, Van Schoubroeck D, Landolfo C, Installe AJ, Guerriero S, Exacoustos C, Gordts S, Benacerraf B, D'Hooghe T, De Moor B, Brolmann H, Goldstein S, Epstein E, Bourne T, Timmerman D. Terms, definitions and measurements to describe sonographic features of myometrium and uterine masses: a consensus opinion from the Morphological Uterus Sonographic Assessment (MUSA) group. Ultrasound Obstet Gynecol. 2015 Sep;46(3):284-98. doi: 10.1002/uog.14806. Epub 2015 Aug 10. PMID 25652685
- [Background] Richtarova A, Boudova B, Dundr P, Lisa Z, Hlinecka K, Zizka Z, Fruhauf F, Kuzel D, Slama J, Mara M. Uterine smooth muscle tumors with uncertain malignant potential: analysis following fertility-saving procedures. Int J Gynecol Cancer. 2023 May 1;33(5):701-706. doi: 10.1136/ijgc-2022-004038. PMID 36898699
- [Background] Giuliani E, As-Sanie S, Marsh EE. Epidemiology and management of uterine fibroids. Int J Gynaecol Obstet. 2020 Apr;149(1):3-9. doi: 10.1002/ijgo.13102. Epub 2020 Feb 17. PMID 31960950
- [Background] Stewart EA, Cookson CL, Gandolfo RA, Schulze-Rath R. Epidemiology of uterine fibroids: a systematic review. BJOG. 2017 Sep;124(10):1501-1512. doi: 10.1111/1471-0528.14640. Epub 2017 May 13. PMID 28296146
- [Result] Stukan M, Rutkowski P, Smadja J, Bonvalot S. Ultrasound-Guided Trans-Uterine Cavity Core Needle Biopsy of Uterine Myometrial Tumors to Differentiate Sarcoma from a Benign Lesion-Description of the Method and Review of the Literature. Diagnostics (Basel). 2022 May 29;12(6):1348. doi: 10.3390/diagnostics12061348. PMID 35741158